CLINICAL TRIAL: NCT03470129
Title: Klinische Bewährung Zweier Fissurenversiegler
Brief Title: Clinical Performance of Two Fissure Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Helioseal F Plus
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Caries Pit and Fissure Limited to Enamel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Helioseal F (Active Comparator): fissure sealing with the conventional product
  Interventions: Device: fissure sealing
- Helioseal F Plus (Experimental): fissure sealing with the new product
  Interventions: Device: fissure sealing

INTERVENTIONS:
Device: fissure sealing — sealing of occlusal fissures with either the conventional sealant, Helioseal F, or the new sealant, Helioseal F Plus, which provides an additional feature and an improved formulation

SUMMARY:
Comparison of the retention of a new fissure sealant (Helioseal F Plus) and a fissure sealant that has been on the market for years in children

ELIGIBILITY:
Inclusion Criteria:

participants

* ASA Status 1
* all dentinal lesions are restored
* consent of parents and patient
* instruction and demonstration of oral hygiene

teeth:

* first and second molars of the permanent dentition
* healthy teeth without caries
* molars with primary lesions

Exclusion Criteria:

participants

* no consent
* allergies to methacrylates or other ingredients of dental products

teeth:

* molars with occlusal cavities (UniViSS score occlusal > M)
* Molars with untreated dentinal lesions
* premolars, incisors, deciduous teeth
* teeth with huge occlusal restorations
* hypomineralized teeth or other defects

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Prof. Jan Kühnisch, München, Bavaria, Germany
- Zahnarztpraxis Graeser, Wädenswil, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment phase took place at both study sites from September 2018 to March 2019.
Units Other Than Participants: Sealants
Period: Overall Study
Arm/Group | Helioseal F | Helioseal F Plus
Started | 92; 164 Sealants | 92; 164 Sealants
12 Month | 85; 152 Sealants | 85; 153 Sealants
24 Month | 82; 148 Sealants | 82; 149 Sealants
Completed | 76; 134 Sealants | 76; 131 Sealants
Not Completed | 16; 30 Sealants | 16; 33 Sealants

BASELINE CHARACTERISTICS:
Population: Split-Mouth Design: Every patient receives both treatments.
Units Other Than Participants: Sealants
Groups:
- Total: Total of all reporting groups
Arm/Group | Helioseal F | Helioseal F Plus | Total
Number analyzed (Participants) | 92 | 92 | 92
Number analyzed (Sealants) | 164 | 164 | 328
Age, Customized [Number; unit: Participants]
  5-18 years | 92 | 92 | 92
Sex/Gender, Customized [Number; unit: participants]
  Female | 51 | 51 | 51
  Male | 41 | 41 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants] — Population: Herein, the participants
  participants
    Switzerland | 41 | 41 | 41
    Germany | 51 | 51 | 51

OUTCOME MEASURES:

1. Primary Outcome: Retention of the Sealant
Description: grade of retention is evaluated as 0 - no fissure sealant left/present 1 complete retention 2 minimal loss of sealant (max one third) 3: central retention of the sealant, 4: almost complete loss of the sealant - less than one third is left
Time Frame: 7-28 days
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 92 | 92
Number analyzed (Sealants) | 164 | 164
Sealants
  0 - no fissure sealant left/present | 0 | 0
  1 complete retention | 164 | 164
  2 minimal loss of sealant (max one third) | 0 | 0
  3: central retention of the sealant, | 0 | 0
  4: almost complete loss of the sealant - less than one third is left | 0 | 0

2. Primary Outcome: Retention of Sealant
Description: as for outcome 1
Time Frame: 12 months
Population: One Sealant of Helioseal F could not be examined due to an orthodontic bite device.
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 85 | 85
Number analyzed (Sealants) | 152 | 153
Sealants
  0 - no fissure sealant left/present | 2 | 2
  1 complete retention | 111 | 116
  2 minimal loss of sealant (max one third) | 24 | 21
  3: central retention of the sealant | 13 | 6
  4: almost complete loss of the sealant - less than one third is left | 2 | 8

3. Primary Outcome: Retention of Sealant
Description: as for outcome 1
Time Frame: 24 months
Population: One Sealant of Helioseal F could not be examined due to an orthodontic bite device.
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 82 | 82
Number analyzed (Sealants) | 148 | 149
Sealants
  0 - no fissure sealant left/present | 0 | 2
  1 complete retention | 100 | 101
  2 minimal loss of sealant (max one third) | 28 | 27
  3: central retention of the sealant | 14 | 11
  4: almost complete loss of the sealant - less than one third is left | 6 | 8

4. Primary Outcome: Retention of Sealant
Description: as for outcome 1
Time Frame: 36 months
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 76 | 76
Number analyzed (Sealants) | 134 | 131
Sealants
  0 - no fissure sealant left/present | 0 | 0
  1 complete retention | 84 | 81
  2 minimal loss of sealant (max one third) | 29 | 26
  3: central retention of the sealant | 15 | 12
  4: almost complete loss of the sealant - less than one third is left | 6 | 12

5. Secondary Outcome: Caries
Description: evaluation of the presence of carious lesions according to UniViSS 2.0
Time Frame: 7-28 days
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 92 | 92
Number analyzed (Sealants) | 164 | 164
Sealants
  No Caries | 164 | 164
  Non-cavitated caries | 0 | 0
  Cavitated caries | 0 | 0

6. Secondary Outcome: Caries
Description: evaluation of the presence of carious lesions according to UniViSS 2.0
Time Frame: 12 months
Population: One Sealant of Helioseal F could not be examined due to an orthodontic bite device.
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 85 | 85
Number analyzed (Sealants) | 152 | 153
Sealants
  No caries | 151 | 151
  Non-cavitated caries | 1 | 2
  Cavitated caries | 0 | 0

7. Secondary Outcome: Caries
Description: evaluation of the presence of carious lesions according to UniViSS 2.0
Time Frame: 24 months
Population: One Sealant of Helioseal F could not be examined due to an orthodontic bite device.
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 82 | 82
Number analyzed (Sealants) | 148 | 149
Sealants
  No caries | 146 | 146
  Non-cavitated caries | 2 | 3
  Cavitated caries | 0 | 0

8. Secondary Outcome: Caries
Description: evaluation of the presence of carious lesions according to UniViSS 2.0
Time Frame: 36 months
Measure: Number; unit: Sealants
Units Other Than Participants: Sealants
Arm/Group | Helioseal F | Helioseal F Plus
Number analyzed (Participants) | 76 | 76
Number analyzed (Sealants) | 134 | 131
Sealants
  No caries | 123 | 120
  Non-cavitated caries | 11 | 11
  Cavitated caries | 0 | 0

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Helioseal F | Helioseal F Plus
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/92 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03470129/Prot_SAP_000.pdf